CLINICAL TRIAL: NCT01383343
Title: Phase I Trial of FOLFIRI in Combination With Sorafenib and Bevacizumab in Patients With Advanced Gastrointestinal Malignancies
Brief Title: Sorafenib Tosylate, Bevacizumab, Irinotecan Hydrochloride, Leucovorin Calcium, and Fluorouracil in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02595; NCI-2011-02595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000702751; MC1017; MC1017 (Other: Mayo Clinic); 8877 (Other: CTEP); P30CA015083 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH)
Record Dates: First submitted 2011-06-25; First posted 2011-06-28 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Recurrent Colon Carcinoma; Recurrent Rectal Carcinoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Fluorouracil; dehydroftorafur; Irinotecan; Leucovorin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (FOLFIRI and bevacizumab) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes on day 1, leucovorin calcium IV over 2 hours on day 1, fluorouracil IV continuously over 46 hours on days 1-2, bevacizumab IV over 30-90 minutes on day 1, and sorafenib tosylate PO QD or BID on days 3-6 and 10-13*. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Fluorouracil; Drug: Irinotecan Hydrochloride; Drug: Leucovorin Calcium; Drug: Sorafenib Tosylate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar FKB238; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase I trial studies the side effects and best dose of sorafenib tosylate when given together with bevacizumab, irinotecan hydrochloride, leucovorin calcium, and fluorouracil in treating patients with colorectal cancer that has spread to other parts of the body. Drugs used in chemotherapy, such as irinotecan hydrochloride, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Sorafenib tosylate and bevacizumab may also block tumor growth in different ways by targeting certain cells. Giving sorafenib tosylate and bevacizumab together with combination chemotherapy may be a better treatment for colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose of the combination of irinotecan hydrochloride, leucovorin calcium, and fluorouracil (FOLFIRI) plus sorafenib (sorafenib tosylate) plus bevacizumab.

SECONDARY OBJECTIVES:

I. To assess the safety of FOLFIRI plus sorafenib plus bevacizumab. II. To assess the feasibility of the proposed combination. III. To evaluate the response rate and identify any activity of the proposed combination.

OUTLINE: This is a dose-escalation study of sorafenib tosylate followed by a cohort study. (Cohort study cancelled as of March 25, 2014)

Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes on day 1, leucovorin calcium IV over 2 hours on day 1, fluorouracil IV continuously over 46 hours on days 1-2, bevacizumab IV over 30-90 minutes on day 1, and sorafenib tosylate orally (PO) once (QD) or twice daily (BID) on days 3-6 and 10-13*. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients may also receive sorafenib tosylate on days 7 and 14.

After completion of study therapy, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* This trial is intended for gastrointestinal malignancies appropriate for irinotecan-based therapy; histologic proof of cancer that is now unresectable; if prior therapy was received, patients must have shown progressive disease during prior treatment or within 6 months of their most recent therapy
* Measurable disease or non-measurable disease
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelet (PLT) >= 100,000/uL
* Hemoglobin (Hgb) >= 9.0 gm/dL
* Total bilirubin =< upper limit of normal (ULN)
* Alkaline phosphatase =< 3 x ULN
* Aspartate aminotransferase (AST) =< 3 x ULN OR AST =< 5 x ULN if liver involvement
* International normalized ratio (INR) < 1.5 unless patients are receiving anti-coagulation therapy; patients receiving anti-coagulation therapy with an agent such as warfarin or heparin are allowed to participate if INR =< 3.0
* Urine protein creatinine (UPC) ratio < 1 or urine dipstick < 2+

  * NOTE: urine protein must be screened by urine analysis for UPC ratio or by dipstick; for UPC ratio >= 1.0, 24-hour urine protein must be obtained and the level should be < 1000 mg
* Creatinine =< 1.5 x ULN
* Calculated creatinine clearance must be >= 45 mL/min using the Cockcroft-Gault formula
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Ability to provide informed consent
* Willing to return to Mayo Clinic for follow up
* Life expectancy >= 84 days (3 months)
* Women of childbearing potential only: negative pregnancy test done =< 7 days prior to registration

Exclusion Criteria:

* Known standard therapy for patient's disease that is potentially curative

Note:

* Prior treatment with irinotecan, 5-fluoruracil or bevacizumab is allowed
* Prior treatment with sorafenib is not allowed

  * Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 100 mmHg on anti-hypertensive medications)
  * Prior history of hypertensive crisis or hypertensive encephalopathy
  * History of myocardial infarction or unstable angina =< 6 months prior to registration or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
  * Heart failure New York Heart Association classification III or IV
  * Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks =< 6 months prior to registration
  * Any hemorrhage/bleeding event > grade 3 =< 4 weeks prior to registration
  * Evidence or history of bleeding diathesis (greater than normal risk of bleeding) or coagulopathy (in the absence of therapeutic anticoagulation); NOTE: patients on full-dose anticoagulants are eligible provided the patient has been on a stable dose for at least 2 weeks of low molecular weight heparin or warfarin and has an INR in the range of 2-3; aspirin doses > 325 mg PO daily are not allowed
  * Active or recent hemoptysis (>= ½ teaspoon of bright red blood per episode) =< 30 days prior to registration
  * Serious, non-healing wound, active ulcer, or untreated bone fracture; NOTE: patients with fractures secondary to metastatic disease are eligible after appropriate radiotherapy
  * Significant vascular disease (e.g., aortic aneurysm, aortic dissection), recent peripheral arterial thrombosis, symptomatic peripheral vascular disease =< 6 months prior to registration
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 6 months prior to registration
  * Major surgical procedures, open biopsy, or significant traumatic injury =< 28 days prior to registration or anticipation of need for major surgical procedure during the course of the study; EXCEPTION: core biopsy or minor surgical procedure, including placement of a vascular access device, =< 7 days prior to registration is allowed
  * Patients taking cytochrome P450 enzyme-inducing antiepileptic drugs =< 4 weeks prior to registration will be excluded (phenytoin, carbamazepine, phenobarbital, rifampin, or St. John's wort)
  * Known or suspected allergy or hypersensitivity to any agent given in the course of this trial
  * Any condition that impairs patient's ability to swallow whole pills
  * Any malabsorption problem
  * Any of the following prior therapies:
* Chemotherapy =< 14 days prior to registration
* Immunotherapy =< 28 days prior to registration
* Radiation therapy =< 28 days prior to registration
* Radiation to > 25% of bone marrow

  * Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
  * Known brain metastasis; NOTE: patients with neurological symptoms must undergo a computed tomography (CT) scan/magnetic resonance imaging (MRI) of the brain to exclude brain metastasis
  * Any of the following:
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

  * Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation)
  * Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
  * Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
  * Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer, including hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of sorafenib tosylate in combination with FOLFIRI and bevacizumab, defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) | 14 days
  Graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Incidence of adverse events of sorafenib tosylate in combination with bevacizumab and FOLFIRI as assessed by NCI CTCAE v 4.0 | Up to 3 months
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Response rate in patients treated with sorafenib tosylate in combination with FOLFIRI and bevacizumab, assessed using Response Evaluation Criteria in Solid Tumors | From the start of the treatment until disease progression/recurrence, assessed up to 3 months
  Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Time to progression | Up to 3 months
Time to treatment failure | Time from registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
Time to until treatment related grade 3+ toxicity assessed via CTC standard toxicity grading | Up to 3 months
  Will be assessed using continuous variables as the outcome measures (primarily nadir). Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Time until any treatment related toxicity evaluated via the ordinal Common Toxicity Criteria (CTC) standard toxicity grading | Up to 3 months
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Time until hematologic nadirs (ANC, platelets, hemoglobin) | Up to 3 months
  Descriptive statistics and simple scatter plots will form the basis of presentation of these data.

CONTACTS AND LOCATIONS:
Overall Officials: Joleen Hubbard, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota